CLINICAL TRIAL: NCT03556566
Title: Open Label, One-arm, 3-month Study of Once-daily Tablet of V3-OVA as Immunotherapy of Ovarian Cancer
Brief Title: Open Label Immunotherapy Trial for Ovarian Cancer
Acronym: V3-OVA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Immunitor LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V3-OVA-01
Record Dates: First submitted 2018-05-26; First posted 2018-06-14 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Ovarian Cancer
Keywords: ovary; ovarian; immunotherapy; cancer
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms

STUDY DESIGN:
Intervention Model Description: Single arm, open label Phase II study in volunteers with ovarian cancer receiving daily dose of one pill of vaccine V3-OVA
Masking Description: no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- V3-OVA treatment arm (Experimental): Oral once daily pill of tableted vaccine (V3-OVA) containing ovarian cancer antigens administered for 3 months in 20 volunteers with ovarian cancer
  Interventions: Biological: Tableted vaccine (V3-OVA) containing ovarian cancer antigens

INTERVENTIONS:
Biological: Tableted vaccine (V3-OVA) containing ovarian cancer antigens — One pill of V3-OVA per day for three months
  Other Names: V3-OVA

SUMMARY:
This Phase II will evaluate a new type of ovarian cancer immunotherapy based on a fundamentally new approach that has been successfully tested in a published clinical study of liver cancer. We will test new tableted preparation, V3-OVA, obtained from hydrolyzed, inactivated blood and tumors of patients with cancer of ovaries. Study will last 3 months, 20 patients will be recruited, given one pill per day for three months. The primary clinical endpoint is effect on tumor size and burden after 3 months. Secondary endpoint will be effect on levels of tumor markers on monthly basis compared to baseline.

DETAILED DESCRIPTION:
Ovarian cancer (OC) - a malignant disease affecting the ovarian tissue - is the sixth most diagnosed cancer among women and causes more deaths than any other cancer of the female reproductive system. For treatment of OC, surgical intervention, chemotherapy, as well as radiation methods are used. Despite treatment, about 70% of patients have a relapse. Many different types of immunotherapy (especially checkpoint inhibitors) of OC being tested, but so far the successes have been insignificant, and serious side effects are frequent and unpredictable. This Phase II will evaluate a new type of ovarian cancer immunotherapy based on a fundamentally new approach that has been successfully tested in a published clinical study of liver cancer. We will test new tableted preparation, V3-OVA, obtained from hydrolyzed, inactivated blood and tumor tissues of patients with cancer of ovaries. Study will last 3 months, 20 patients will be recruited, given one pill per day for three months. The primary clinical endpoint is effect on tumor size and burden after 3 months. Secondary endpoint will be effect on levels of tumor markers on monthly basis compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

Confirmed diagnosis of ovarian cancer Positive for CA125 tumor marker at above normal threshold level -

Exclusion Criteria:

Metastases to other sites

-

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Ovarian cancer is female gynecological cancer
Enrollment: 20 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in tumor size and burden compared to baseline | Monthly for 3 months
  Intravaginal ultrasonography to measure changes in tumor size and burden

SECONDARY OUTCOMES:
Effect on level of serum tumor markers compared to baseline | Monthly for three months
  Commonly measured tumor markers associated with ovarian cancer, primarily CA125, at baseline and at study termination

CONTACTS AND LOCATIONS:
Overall Officials: Aldar Bourinbaiar, PhD, MD/PhD, Study Chair — Immunitor LLC
Locations (1):
- Immunitor LLC, Ulaanbaatar, Mongolia

IPD SHARING:
Plan to Share IPD: No
Data will be shared upon study completion in peer-reviewed publication